CLINICAL TRIAL: NCT04216667
Title: Posterior Wall And Left Atrial Appendage Empiric Electrical Isolation for Non-Paroxysmal Atrial Fibrillation (The PLEA Trial)
Brief Title: Posterior Wall And Left Atrial Appendage Empiric Electrical Isolation for Non-Paroxysmal Atrial Fibrillation
Acronym: PLEA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Montefiore Medical Center (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-10714
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation; Arrhythmia Recurrence; Embolic Stroke; Mortality
MeSH Terms: conditions — Atrial Fibrillation; Embolic Stroke | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: A total of 932 patients will be randomized with equal allocation to one of four treatment groups. This sample size provides 90% power to detect pairwise differences in response rates between groups ranging from 0.12 to 0.15 based on two-tailed 0.05 level intention to treat chi-squared tests. Specifically, the response rates under the alternative upon which sample size is determined are 0.45, 0.60, 0.75, 0.87 for PVI alone, PVI + PWI, PVI + PWI + LAAEI and PVI + PWI + LAAEI + CSI respectively.
Who Masked: Participant, Outcomes Assessor
Masking Description: The nature of the ablation procedures precludes blinding of physicians to patient treatment. However, patients will be blinded to their ablation strategy (single-blind design) and endpoint assessment will be made by blinded adjudicators from an independent core laboratory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PVI (Active Comparator): Pulmonary vein isolation alone will be performed using radiofrequency energy
  Interventions: Procedure: Catheter ablation
- PVI + PWI (Experimental): Pulmonary vein isolation plus posterior wall isolation will be performed using radiofrequency energy
  Interventions: Procedure: Catheter ablation
- PVI + PWI + LAAEI (Experimental): Pulmonary vein isolation plus posterior wall isolation plus left atrial appendage electrical isolation will be performed using radiofrequency energy
  Interventions: Procedure: Catheter ablation
- PVI + PWI + LAAEI + CSI (Experimental): Pulmonary vein isolation plus posterior wall isolation plus left atrial appendage electrical isolation plus coronary sinus isolation will be performed using radiofrequency energy
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Catheter ablation

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of empirical posterior wall isolation (PWI), left atrial appendage electrical isolation (LAAEI) and coronary sinus isolation (CSI) when compared to pulmonary vein isolation (PVI) alone:

* PVI alone,
* PVI + PWI,
* PVI + PWI + LAAEI,
* PVI + PWI + LAAEI + CSI.

DETAILED DESCRIPTION:
The Posterior Wall and/or Left Atrial Appendage Empiric Electrical Isolation for Non-Paroxysmal Atrial Fibrillation (The PLEA Trial) is a prospective multicenter randomized controlled study that has the overall goal of establishing the efficacy and safety of different ablation techniques for patients with persistent and long-standing persistent atrial fibrillation. The PLEA trial is designed to test the hypothesis whether posterior wall isolation (PWI) with pulmonary vein isolation (PVI), PWI plus left atrial appendage electrical isolation (LAAEI) with PVI and PWI plus LAAEI plus coronary sinus isolation (CSI) with PVI is superior to the standard approach alone (i.e. PVI alone) in decreasing the incidence of the composite endpoint of all-cause mortality and all-atrial arrhythmia recurrences.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or greater
4. In good general health as evidenced by medical history and diagnosed with symptomatic persistent AF or long-standing persistent AF.

   1. Persistent AF will be defined as a sustained episode lasting > 7 days and less than 1 year.
   2. Long-standing persistent AF will be defined as a sustained episode lasting more than 1 year and less than 10 years.
   3. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, left ventricular dysfunction, or other symptoms, or any combination of the above.
5. At least one episode of persistent AF must have been documented by ECG, Holter, loop recorder, ziopatch, telemetry, trans telephonic monitoring (TTM), or implantable device within last 10 years of enrollment in this investigation.
6. Patients undergoing first time procedure for AF.

Exclusion Criteria:

1. Patients with paroxysmal AF.

   • Paroxysmal AF will be defined as a sustained episode lasting < 7 days (either terminated spontaneously or with pharmacological or electrical cardioversion.
2. Reversible causes of AF.
3. Patients with contraindications to systemic anticoagulation with heparin or coumadin, direct thrombin inhibitor or factor Xa inhibitors.
4. Patients with left atrial size ≥ 75 mm (2D echocardiography, parasternal long axis view)
5. Left atrial or LAA thrombus
6. Patients with severe valvular heart disease or after mitral valve replacement (bioprosthetic or mechanical).
7. Patients with a life expectancy ≤ 24 months
8. CHA2DS2Vasc score of 0 for men and CHA2DS2Vasc score of 1 for women.
9. Patients who are pregnant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Freedom from documented AF/AT/AFL episodes and all-cause mortality after initial procedure | 12 months
  The primary effectiveness endpoint is defined as the freedom from documented AF/AT/AFL episodes (> 30 seconds) and all-cause mortality within 12 months after one ablation procedure without antiarrhythmic medications after blanking period (3 months after ablation) as adjudicated by the independent Core Laboratory.
  Atrial Fibrillation (AF) Atrial Tachycardia (AT) Atrial Flutter (AFL)
A composite of thromboembolic events, myocardial perforation, pulmonary vein stenosis, atrioesophageal fistula, left and right phrenic nerve paralysis, and other serious adverse events within 12 months post-procedure. | 12 months
  The primary safety endpoint is defined as a composite of thromboembolic events, myocardial perforation, pulmonary vein stenosis, atrioesophageal fistula, left and right phrenic nerve paralysis, and other serious adverse events within 12 months post-procedure.

SECONDARY OUTCOMES:
Incidence of peri-procedural and 12-month post procedural complications. | 12, 24 and 60 months
  These complications include: ischemic stroke, pulmonary veins (PVs) stenosis, cardiac perforation, esophageal injury, phrenic nerve paralysis, rehospitalization, and death.
AF/AT/AFL Burden | 12, 24 and 60 months
  Atrial fibrillation (AF), atrial tachycardia (AT) and/or atrial flutter (AFL) burden at 12 months after single and redo procedures
All-cause mortality | 12, 24 and 60 months
  Death from all causes will be assessed
Atrial contractility | 6 months
  Myocardial strain will be used to assess atrial contractility after catheter ablation
Heart failure analysis | 12, 24 and 60 months
  Primary outcome will be assessed base on left ventricular ejection fraction (LVEF)
Cardiovascular hospitalizations | 12, 24 and 60 months
  Cardiovascular hospitalization was characterized by the site principal investigator (PI) and reported as part of the hospitalization case report form.
Procedure duration and fluoroscopy time | Day of Procedure
  These times will be compared amongst groups
Number of repeat procedures | 12 months
  Number of repeat procedures within 12 months after the first ablation procedure
Cost-effectiveness analysis | 12 months
  The CEA will examine the cost of health care resources and health outcomes from the ablation procedure to 1-year postoperatively. The costs will include all health care utilization during this time. Health care utilization, and associated costs, related to the patients' condition, the procedure and adverse events will be the basis of a sensitivity analysis.
Long-term follow-up at 24 and 60 months to evaluate freedom of documented AF/AT/AFL episodes (>30 seconds) and all-cause mortality adjudicated by the Core Laboratory | 24 and 60 months
  Freedom from documented AF/AT/AFL episodes (> 30 seconds) and all-cause mortality within 24 and 60 months after one ablation procedure without antiarrhythmic medications after blanking period (3 months after ablation) as adjudicated by the independent Core Laboratory.
  Atrial Fibrillation (AF) Atrial Tachycardia (AT) Atrial Flutter (AFL)
Freedom from documented AF/AT/AFL episodes (>30 seconds) and all-cause mortality within 12 months after redo ablation procedure. | 12 months
  Freedom from all-atrial arrhythmias recurrence (AF/atrial flutter [AFL]/atrial tachycardia [AT]) (episodes >30 seconds on 12-lead ECG, event monitor, Zio patch, Holter or device interrogation) and all-cause mortality (patients who die before the 12-month assessment or who are too ill to undergo assessment of AF are considered not to have response to treatment) during the evaluation period at 12 months after redo-ablation procedures as adjudicated by the independent Core Laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Romero, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine; Luigi Di Biase, MD, PhD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine; Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Institute and St. David's Medical Center
Locations (16):
- United States (10):
  - Grandview Medical Center, Birmingham, Alabama
  - MarinHealth Medical Center, Larkspur, California
  - University of Colorado, Boulder, Colorado
  - Miami Cardiac & Vascular Institute, Miami, Florida
  - Indiana University, Bloomington, Indiana
  - Montefiore Medical Center, The Bronx, New York
  - WakedMed Heart & Vascular, Raleigh, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Institute, Austin, Texas
  - Baylor Heart Clinic, Houston, Texas
- Instituto Cardiovascular Adventista, Buenos Aires, Argentina
- Incor - HCFMUSP, São Paulo, Brazil
- University CES, Medellín, Antioquia, Colombia
- Cardioangiologisches Centrum Bethanien, Frankfurt, Germany
- Hospital Santa Cruz, Lisbon, Portugal
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero J, Michaud GF, Avendano R, Briceno DF, Kumar S, Carlos Diaz J, Mohanty S, Trivedi C, Gianni C, Della Rocca D, Proietti R, Perrotta L, Bordignon S, Chun JKR, Schmidt B, Garcia M, Natale A, Di Biase L. Benefit of left atrial appendage electrical isolation for persistent and long-standing persistent atrial fibrillation: a systematic review and meta-analysis. Europace. 2018 Aug 1;20(8):1268-1278. doi: 10.1093/europace/eux372. PMID 29342299
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. Europace. 2018 Jan 1;20(1):157-208. doi: 10.1093/europace/eux275. No abstract available. PMID 29016841
- [Background] Di Biase L, Burkhardt JD, Mohanty P, Mohanty S, Sanchez JE, Trivedi C, Gunes M, Gokoglan Y, Gianni C, Horton RP, Themistoclakis S, Gallinghouse GJ, Bailey S, Zagrodzky JD, Hongo RH, Beheiry S, Santangeli P, Casella M, Dello Russo A, Al-Ahmad A, Hranitzky P, Lakkireddy D, Tondo C, Natale A. Left Atrial Appendage Isolation in Patients With Longstanding Persistent AF Undergoing Catheter Ablation: BELIEF Trial. J Am Coll Cardiol. 2016 Nov 1;68(18):1929-1940. doi: 10.1016/j.jacc.2016.07.770. PMID 27788847
- [Background] Ludka L. [Fasting during childbirth]. Katilolehti. 1988 Sep;93(6):25-8. No abstract available. Finnish. PMID 3210508
- [Background] Allessie MA, de Groot NM, Houben RP, Schotten U, Boersma E, Smeets JL, Crijns HJ. Electropathological substrate of long-standing persistent atrial fibrillation in patients with structural heart disease: longitudinal dissociation. Circ Arrhythm Electrophysiol. 2010 Dec;3(6):606-15. doi: 10.1161/CIRCEP.109.910125. Epub 2010 Aug 18. PMID 20719881
- [Background] Brooks AG, Stiles MK, Laborderie J, Lau DH, Kuklik P, Shipp NJ, Hsu LF, Sanders P. Outcomes of long-standing persistent atrial fibrillation ablation: a systematic review. Heart Rhythm. 2010 Jun;7(6):835-46. doi: 10.1016/j.hrthm.2010.01.017. Epub 2010 Jan 22. PMID 20206320
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Lim HS, Hocini M, Dubois R, Denis A, Derval N, Zellerhoff S, Yamashita S, Berte B, Mahida S, Komatsu Y, Daly M, Jesel L, Pomier C, Meillet V, Amraoui S, Shah AJ, Cochet H, Sacher F, Jais P, Haissaguerre M. Complexity and Distribution of Drivers in Relation to Duration of Persistent Atrial Fibrillation. J Am Coll Cardiol. 2017 Mar 14;69(10):1257-1269. doi: 10.1016/j.jacc.2017.01.014. PMID 28279292
- [Background] Bai R, Di Biase L, Mohanty P, Trivedi C, Dello Russo A, Themistoclakis S, Casella M, Santarelli P, Fassini G, Santangeli P, Mohanty S, Rossillo A, Pelargonio G, Horton R, Sanchez J, Gallinghouse J, Burkhardt JD, Ma CS, Tondo C, Natale A. Proven isolation of the pulmonary vein antrum with or without left atrial posterior wall isolation in patients with persistent atrial fibrillation. Heart Rhythm. 2016 Jan;13(1):132-40. doi: 10.1016/j.hrthm.2015.08.019. Epub 2015 Aug 13. PMID 26277862
- [Background] Tamborero D, Mont L, Berruezo A, Matiello M, Benito B, Sitges M, Vidal B, de Caralt TM, Perea RJ, Vatasescu R, Brugada J. Left atrial posterior wall isolation does not improve the outcome of circumferential pulmonary vein ablation for atrial fibrillation: a prospective randomized study. Circ Arrhythm Electrophysiol. 2009 Feb;2(1):35-40. doi: 10.1161/CIRCEP.108.797944. Epub 2008 Dec 3. PMID 19808442
- [Background] Lim TW, Koay CH, See VA, McCall R, Chik W, Zecchin R, Byth K, Seow SC, Thomas L, Ross DL, Thomas SP. Single-ring posterior left atrial (box) isolation results in a different mode of recurrence compared with wide antral pulmonary vein isolation on long-term follow-up: longer atrial fibrillation-free survival time but similar survival time free of any atrial arrhythmia. Circ Arrhythm Electrophysiol. 2012 Oct;5(5):968-77. doi: 10.1161/CIRCEP.111.970293. Epub 2012 Sep 12. PMID 22972873
- [Background] Aryana A, Baker JH, Espinosa Ginic MA, Pujara DK, Bowers MR, O'Neill PG, Ellenbogen KA, Di Biase L, d'Avila A, Natale A. Posterior wall isolation using the cryoballoon in conjunction with pulmonary vein ablation is superior to pulmonary vein isolation alone in patients with persistent atrial fibrillation: A multicenter experience. Heart Rhythm. 2018 Aug;15(8):1121-1129. doi: 10.1016/j.hrthm.2018.05.014. PMID 30060879
- [Background] Di Biase L, Burkhardt JD, Mohanty P, Sanchez J, Mohanty S, Horton R, Gallinghouse GJ, Bailey SM, Zagrodzky JD, Santangeli P, Hao S, Hongo R, Beheiry S, Themistoclakis S, Bonso A, Rossillo A, Corrado A, Raviele A, Al-Ahmad A, Wang P, Cummings JE, Schweikert RA, Pelargonio G, Dello Russo A, Casella M, Santarelli P, Lewis WR, Natale A. Left atrial appendage: an underrecognized trigger site of atrial fibrillation. Circulation. 2010 Jul 13;122(2):109-18. doi: 10.1161/CIRCULATIONAHA.109.928903. Epub 2010 Jul 6. PMID 20606120
- [Background] Hocini M, Shah AJ, Nault I, Sanders P, Wright M, Narayan SM, Takahashi Y, Jais P, Matsuo S, Knecht S, Sacher F, Lim KT, Clementy J, Haissaguerre M. Localized reentry within the left atrial appendage: arrhythmogenic role in patients undergoing ablation of persistent atrial fibrillation. Heart Rhythm. 2011 Dec;8(12):1853-61. doi: 10.1016/j.hrthm.2011.07.013. Epub 2011 Jul 12. PMID 21762673
- [Background] Panikker S, Jarman JW, Virmani R, Kutys R, Haldar S, Lim E, Butcher C, Khan H, Mantziari L, Nicol E, Foran JP, Markides V, Wong T. Left Atrial Appendage Electrical Isolation and Concomitant Device Occlusion to Treat Persistent Atrial Fibrillation: A First-in-Human Safety, Feasibility, and Efficacy Study. Circ Arrhythm Electrophysiol. 2016 Jul;9(7):e003710. doi: 10.1161/CIRCEP.115.003710. PMID 27406602
- [Background] Yorgun H, Canpolat U, Kocyigit D, Coteli C, Evranos B, Aytemir K. Left atrial appendage isolation in addition to pulmonary vein isolation in persistent atrial fibrillation: one-year clinical outcome after cryoballoon-based ablation. Europace. 2017 May 1;19(5):758-768. doi: 10.1093/europace/eux005. PMID 28340073
- [Background] Lakkireddy D, Sridhar Mahankali A, Kanmanthareddy A, Lee R, Badhwar N, Bartus K, Atkins D, Bommana S, Cheng J, Rasekh A, Di Biase L, Natale A, Nath J, Ferrell R, Earnest M, Reddy YM. Left Atrial Appendage Ligation and Ablation for Persistent Atrial Fibrillation: The LAALA-AF Registry. JACC Clin Electrophysiol. 2015 Jun;1(3):153-160. doi: 10.1016/j.jacep.2015.04.006. Epub 2015 Apr 30. PMID 29759358
- [Background] Romero J, Natale A, Di Biase L. Left atrial appendage empirical electrical isolation for persistent atrial fibrillation: time for a change in practice. Europace. 2017 May 1;19(5):699-702. doi: 10.1093/europace/eux050. No abstract available. PMID 28402461
- [Background] Heeger CH, Rillig A, Geisler D, Wohlmuth P, Fink T, Mathew S, Tilz RR, Reissmann B, Lemes C, Maurer T, Santoro F, Inaba O, Sohns C, Huang Y, Alessandrini H, Dotz I, Schluter M, Metzner A, Kuck KH, Ouyang F. Left Atrial Appendage Isolation in Patients Not Responding to Pulmonary Vein Isolation. Circulation. 2019 Jan 29;139(5):712-715. doi: 10.1161/CIRCULATIONAHA.118.037451. No abstract available. PMID 30689416
- [Derived] Diaz JC, Canas F, Duque M, Aristizabal J, Nino C, Bastidas O, Marin J, Rivera E, Hoyos C, Matos C, Peralta A, Martin DT, Romero J. Assisted reality device to guide cardiac implantable device programming in distant rural areas. J Cardiovasc Electrophysiol. 2023 Mar;34(3):497-501. doi: 10.1111/jce.15815. Epub 2023 Jan 22. PMID 36640437
- [Derived] Osorio J, Varley A, Kreidieh O, Godfrey B, Schrappe G, Rajendra A, Silverstein J, Romero J, Rodriguez D, Morales G, Zei P. High-Frequency, Low-Tidal-Volume Mechanical Ventilation Safely Improves Catheter Stability and Procedural Efficiency During Radiofrequency Ablation of Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2022 Apr;15(4):e010722. doi: 10.1161/CIRCEP.121.010722. Epub 2022 Mar 25. No abstract available. PMID 35333095